CLINICAL TRIAL: NCT05430074
Title: Treatment of Paediatric Supracondylar Humeral Fracture With Cast Immobilization: A Randomized Controlled Trial - Hybrid Mesh Versus Fibreglass
Brief Title: HM vs Fibreglass Cast Immbolization for Supracondylar Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Principal Investigator, Kenneth Wong Pak Leung, Consultant, KK Women's and Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIRB Ref: 2022/2409
Record Dates: First submitted 2022-06-16; First posted 2022-06-24 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Pediatric Supracondylar Humeral Fracture
Keywords: Supracondylar humeral fracture; Pediatric fracture; Hybrid mesh cast; Fibreglass cast
MeSH Terms: interventions — Casts, Surgical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HM Cast (Other)
  Interventions: Device: HM Cast
- Fibreglass Cast (Other)
  Interventions: Device: Fibreglass Cast

INTERVENTIONS:
Device: HM Cast — Subjects assigned to this arm will be treated via cast immobilisation with the use of HM casts.
  Arms: HM Cast
Device: Fibreglass Cast — Subjects assigned to this arm will be treated via cast immobilisation with the use of Fibreglass casts.
  Arms: Fibreglass Cast

SUMMARY:
Supracondylar humeral fractures are the most common elbow fractures in children and cast immobilization continues to remain as the recommended treatment for modified Gartland's classification Type I and Type IIa injuries. Apart from plaster of Paris and fibreglass casts, the use of waterproof, tubular hybrid mesh (HM) casts have been gaining traction for cast immobilization. Although the use of HM cast has been reported to have similar clinical outcomes and overall patient satisfaction scores to the fibreglass cast, the results of the recent studies are only limited and generalizable only to paediatric distal radius fractures.

As the application method of HM and fibreglass casts are fundamentally different, it has not been reported if the difference in application duration between the cast materials is significant and its potential implications in outpatient clinic operation.

Hence, through a randomized controlled trial, this study primarily aims to investigate if the clinical outcomes, patient satisfaction and duration of cast application with the HM casts would be comparable with fibreglass casts in children with supracondylar humeral fractures.

Through this study, the investigators hope to evaluate the advantages and disadvantages of the respective casting material which may better aid physicians in deciding a more appropriate cast material for treating paediatric supracondylar humeral fractures with cast immobilization and the implications of casting duration on clinic operations.

ELIGIBILITY:
Inclusion Criteria:

* First Presentation of Supracondylar humeral fracture (Type I and IIa modified Gartland's classification)

Exclusion Criteria:

* Prior treatment of supracondylar humeral fracture
* Previous elbow injuries
* Open fractures
* Polytrauma
* Neurovascular injuries

Ages: 0 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 79 (Actual)
Dates: Start 2022-08-16 (Actual); Primary Completion 2022-11-28 (Actual); Study Completion 2022-11-28 (Actual)

PRIMARY OUTCOMES:
Clinical Outcome - Loss of Reduction | 4 weeks post-casting
  Based on the radiographs taken 4 weeks after casting, the Baumann's angle will used to assess for any loss of reduction.
Comfort and Overall Satisfaction | 4 weeks post-casting
  Through a questionnaire, the patients and their parents will be asked to rate the patients' experience on adaptability, weight of the cast, itch, heat, sweatiness, smell, comfort and overall satisfaction. For each question, on the scales of 1 to 5, the rating of 1 would designate as the least desirable option and the rating of 5 being the most desirable option.
Presence of Skin Rash | 4 weeks post-casting
  The presence of skin rash will be assessed by the study team member upon cast removal.

SECONDARY OUTCOMES:
Duration of Cast Application | During Procedure (Cast Application - First Visit)
  The duration of each cast application with the respective cast materials will be recorded and analysed.

OTHER OUTCOMES:
Water Contact (For HM casts only) | 4 weeks post-casting
  Through a questionnaire, patients with HM casts will be asked if they had wetted their casts during showers/baths and if they had participated in any water activities (such as swimming or visits to the waterparks).
Duration and Intensity of Pain | 4 weeks post-casting
  Patients will be assessed based on the duration and intensity of pain, and the duration of painkillers used. The intensity of the pain will be assessed via the Faces Pain Scale - Revised, which is a validated self-reporting measure for children to score their pain on rating from 0 to 10, with 0 being "No pain" and 10 being "Very much pain".

CONTACTS AND LOCATIONS:
Locations (1):
- KK Women's and Children Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No